CLINICAL TRIAL: NCT04368338
Title: Use of Lung Ultrasound in Patients Suspected of COVID-19 Infection in the Emergency Room
Brief Title: Lung Ultrasound to Diagnose COVID-19
Acronym: COVILUS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2020_843_0030
Record Dates: First submitted 2020-04-28; First posted 2020-04-29 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Covid-19; Lung Ultrasound; Respiratory Complication
Keywords: Covid-19; lung ultrasound; Respiratory Complication
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Nucleic Acid Testing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: COVID-19 RT-PCR — Polymerase chain reaction tests after reverse transcription for the detection of viral Covid-19 RNA (RT-PCR)
Procedure: lung ultrasound — lung ultrasound is standard practice to diagnose acute respiratory failure in Emergency room

SUMMARY:
Covid-19 (English acronym meaning coronavirus disease 2019) is an emerging infectious disease caused by a strain of coronavirus called SARS-CoV-2. The current pandemic has resulted in a significant number of admissions in the emergency room (ER) due to suspicion of COVID-19 infection. Use of lung ultrasound is standard practice to diagnose acute respiratory failure in ER. Recently, typical lung ultrasonographic characteristics of COVID-19 disease has been described. During the COVID-19 pandemic, the use of this tool could be of interest in order to allow an early, simple and reliable triage in patients with suspected COVID-19 infection admitted in ER. In addition, the visualization of early signs in specific areas could be a predictive marker of the severity of the disease. The objective of this project will be to study the association between the signs on lung ultrasound and the result of RT-PCR in patients with suspected COVID-19 infection in the ER.

ELIGIBILITY:
Inclusion Criteria:

* patients admitted to Emergency Room for suspicion of COVID-19 infection with has a SARS-CoV-2 RT-PCR test and for whom the emergency doctor decide to perform a lung ultrasound

Exclusion Criteria:

* patients < 18 years of age or under guardianship or curators,
* pregnancy
* poor echogenicity due to the presence of an acoustic barrier (pneumothorax, subcutaneous emphysema, etc.)
* patients with a suspected or proven acute lung disease (pneumonitis, acute respiratory distress syndrome (ARDS))
* chronic interstitial lung disease
* patients who will refuse to give their consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to Emergency Room (ER) for suspicion of COVID-19 infection who has a SARS-CoV-2 RT-PCR test and for whom the emergency doctor decide to perform a lung ultrasound as part of the BLUE protocol.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-04-28 (Actual); Primary Completion 2021-01-28 (Actual); Study Completion 2021-07-20 (Actual)

PRIMARY OUTCOMES:
Lung ultrasound/biological correlation research modulating the severity of Covid-19 disease | 6 months
  Polymerase chain reaction tests after reverse transcription for the detection of covid-19 viral RNA will be done as biological test.

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Bar, MD, Principal Investigator — CHU Amiens
Locations (1):
- BAR, Amiens, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bar S, Lecourtois A, Diouf M, Goldberg E, Bourbon C, Arnaud E, Domisse L, Dupont H, Gosset P. The association of lung ultrasound images with COVID-19 infection in an emergency room cohort. Anaesthesia. 2020 Dec;75(12):1620-1625. doi: 10.1111/anae.15175. Epub 2020 Jul 1. PMID 32520406